CLINICAL TRIAL: NCT04366661
Title: Iraqi Trial for Lung Cancer Screening
Acronym: ITLUCAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Oncology Teaching Hospital, Baghdad (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: OTH267
Record Dates: First submitted 2020-04-22; First posted 2020-04-29 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Lung Cancer
Keywords: smoking; envirumental polution
MeSH Terms: conditions — Lung Neoplasms; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- screening (Experimental): Participants undergo low dose CT of the chest
  Interventions: Diagnostic Test: low dose CT

INTERVENTIONS:
Diagnostic Test: low dose CT — Invited participants from institutes exposed to a high level of smoke pollution such as employees of Transport and Oil Ministries are inquired for their personal history of cigarette smoking then subjected to low dose CT

SUMMARY:
Lung cancer is a global problem. Worldwide, 1.2 million people die of lung cancer each year. In Iraq, lung cancer is the most common malignancy after breast cancer and the leading cause of cancer-related death. Tobacco smoking plays a major role in lung cancer; it is reported in 85-90% of lung cancer patients yet environmental tobacco smoke, environmental and domestic air pollution, work-related risk factors, radon exposure, and viruses may also have an impact on lung cancer incidence rates. Early detection of the disease before patients develop symptoms considers the best way to improve patient outcomes. IT LUCAS is designed to evaluate the utility of low-dose computed tomography (LDCT) screening in early detection and management of lung cancer in high-risk people.

DETAILED DESCRIPTION:
Background Lung cancer is a global problem. Worldwide, 1.2 million people die of lung cancer each year. In Iraq, lung cancer is the most common malignancy after breast cancer and the leading cause of cancer-related death. Tobacco smoking plays a major role in lung cancer; it is reported in 85-90% of lung cancer patients yet environmental tobacco smoke, environmental and domestic air pollution, work-related risk factors, radon exposure, and viruses may also have an impact on lung cancer incidence rates. Early detection of the disease before patients develop symptoms considers the best way to improve patient outcomes. Screening for lung cancer using low dose computed tomography (LDCT) has been the subject of research studies since the 1990s. It has been reported to be superior to CXR and septum cytology for small tumors detection.

Aim of the study IT LUCAS is designed to evaluate the utility of LDCT screening in early detection and management of lung cancer in high-risk people in Iraq.

Study design 500 healthy participants aged 50-75 years with a history of smoking of at least 30 pack year of smoking were recruited from Ministries of Oil and Transport. They were offered Low dose CT of the chest. Nodules with suspicious (Lung RADs 4A or 4B) findings were classified as positive and referred to the Respiratory Department for further workup and biopsy. Nodules with Lung RADS 3 features are reviewed after 6 months while those with Lung RADS 2 offered a LDCT after 12 months.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* aged between 50 and 75
* smokers or ex-smoker
* tobacco exposure of more than 30 pack-years

Exclusion Criteria:

* History of cancer within the last 5 years other than non-melanoma skin cancer or carcinoma in situ,
* heart or respiratory severe co-morbidity with contraindications to thoracoscopy

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
The efficacy of LD CT in lung cancer screening | 2 years
  The number of lung nodules with Lung RADS 4A, 4B and 4X, cancer predictive value and false-positive value

SECONDARY OUTCOMES:
noncancerous lung lesions | 2 years
  the number of nodules with Lung RADS 2 and 3 features

CONTACTS AND LOCATIONS:
Overall Officials: Enam A Khalil, Principal Investigator — Oncology Teaching Hospital
Locations (1):
- Oncology Teaching Hospital, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Iraqi Cancer Rigistry — http://moh.gov.iq/upload/upfile/ar/882.pdf